CLINICAL TRIAL: NCT01138293
Title: Electronic Health Technology for Assessment of Physical Activity and Eating Habits in Children and Adolescents Who Are Overweight and Those With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEDIGREIF Inselklinik Heringsdorf (Network)
Collaborators: Fraunhofer Institut für Graphische Datenverarbeitung (IGD), Rostock, Germany (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDIGREIF 001
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Overweight; Obesity
Keywords: differences between patients´ self-assessment and objective perception of physical activity and eating habits
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- motion sensor integrated in a mobile phone (Experimental): A motion sensor integrated in a mobile phone. The system analyses kind, intensity and duration of physical activity and eating habits.
  Interventions: Device: motion detection with a motion sensor

INTERVENTIONS:
Device: motion detection with a motion sensor — To asses physical activity and eating habits electronic health technology was used (Fraunhofer-Institute). The system consists in a motion sensor integrated in a mobile phone (DiaTrace). The system analyses kind, intensity and duration of physical activity and eating habits.

SUMMARY:
Aims: During the last decades overweight/obesity has increased markedly. They are associated with a high risk for diabetes and death. Effective intervention is mandatory. Following participation in treatment programmes children/adolescents often fail to reach sufficient long-term weight reduction. The present trial aims to integrate telemedical support in therapy to improve long term outcome.

Methods: All children/adolescents with overweight/obesity were included (n=66,age 13.9±2.6 years, body mass index [BMI] 31.2±5.4kg/m², body mass index standard deviation score [BMI-SDS] 2.41±0.6) admitted to our hospital 04-03/2009. To asses physical activity and eating habits electronic health technology was used (Fraunhofer-Institute). The system consists in a motion sensor integrated in a mobile phone(DiaTrace). The system analyses kind, intensity and duration of physical activity and eating habits.

ELIGIBILITY:
Inclusion Criteria:

* All children/adolescents with overweight/obesity were included admitted to our hospital

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MEDIGREIF Inselklinik Heringsdorf GmbH, Haus Gothensee, Heringsdorf, Germany